CLINICAL TRIAL: NCT00193037
Title: A Phase II Randomized Crossover Study Doxorubicin HCI Liposome Injection Versus Weekly Docetaxel in Patients First Relapse Metastatic Breast Cancer
Brief Title: Doxorubicin HCI Liposome Injection Versus Weekly Docetaxel in Patients First Relapse Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Ortho Biotech, Inc. (Industry); Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 43
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2013-07-19 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposomal Doxorubicin (Experimental): Liposomal doxorubicin 40 mg/m2 by 1 hour IV infusion repeated every 28 days.
  Interventions: Drug: Liposomal Doxorubicin
- Docetaxel (Experimental): Weekly docetaxel 36 mg/m2 by 30 minute IV infusion on days 1, 8, and 15 of the 28 day cycle
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Liposomal Doxorubicin — Liposomal Doxorubicin
  Other Names: Doxil
  Arms: Liposomal Doxorubicin
Drug: Docetaxel — Docetaxel
  Other Names: Taxotere
  Arms: Docetaxel

SUMMARY:
The efficacy of single agent liposomal doxorubicin as compared to single agent docetaxel will be evaluated as first line treatment in metastatic breast cancer patients, with subsequent crossover to the opposite arm at disease progression or patient intolerance. We will explore this as well as any possible cross resistance between these two agents.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be randomly assigned to one of two treatment arms:

* Liposomal Doxorubicin
* Docetaxel

For ever 2 patients treated, 1 will receive treatment A (Liposomal Doxorubicin) and 1 will receive treatment B (Docetaxel). Patients demonstrating progression on either ARM will be eligible for cross over to treatment in the other ARM, provided patient still meets the eligibility laboratory and performance status criteria. The study is not blinded so both the patient and the doctor will know which treatment has been assigned.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Metastatic breast cancer confirmed by biopsy
* Prior adjuvant/neoadjuvant treatment allowed
* Measurable disease
* Able to perform activities of daily living with minimal assistance
* Age 18 years or older
* Adequate bone marrow, liver and kidney function
* Normal heart function
* Written informed consent

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Pre-existing moderate peripheral neuropathy
* History of significant heart disease
* Meningeal metastases.
* Prior chemotherapy for metastatic breast cancer
* No measurable disease (including bone only, pleural effusions, etc.)
* Receiving Herceptin therapy.
* Women who are pregnant or lactating.

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2001-02; Primary Completion 2008-12 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, Nashville, Tennessee, United States

REFERENCES:
- [Result] Yardley DA, Burris HA 3rd, Spigel DR, Clark BL, Vazquez E, Shipley D, Barton J, Thompson D, Montes I, Greco FA, Hainsworth JD. A phase II randomized crossover study of liposomal doxorubicin versus weekly docetaxel in the first-line treatment of women with metastatic breast cancer. Clin Breast Cancer. 2009 Nov;9(4):247-52. doi: 10.3816/CBC.2009.n.042. PMID 19933081
- See also: Published article in Clinical Breast Cancer — http://cigjournals.metapress.com/content/h221p3m53r461w57/fulltext.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A -Liposomal Doxorubicin Then Docetaxel: Liposomal doxorubicin (Arm A)
  Liposomal doxorubicin 40 mg/m2 IV day 1 over one hour, repeated q 28 days thru peripheral vein or central venous access. This will define one cycle.
  Patients demonstrating progression on Liposomal Doxorubicin were eligible for cross over to treatment on Docetaxel, provided patient still met the eligibility laboratory and performance status criteria.
- Arm B - Docetaxel Then Liposomal Doxorubicin: Weekly docetaxel 36 mg/m2 IV over 30 minutes on days 1, 8 and 15 followed by one week rest, administered on a q 28 day cycle. This dosing schedule will define one cycle.
  Patients demonstrating progression on Docetaxel were eligible for cross over to treatment on Liposomal Doxorubicin, provided patient still met the eligibility laboratory and performance status criteria.
Period: Randomized Treatment
Arm/Group | Arm A -Liposomal Doxorubicin Then Docetaxel | Arm B - Docetaxel Then Liposomal Doxorubicin
Started | 50 | 52
Completed | 32 | 24
Not Completed | 18 | 28
Period: Crossover Treatment
Arm/Group | Arm A -Liposomal Doxorubicin Then Docetaxel | Arm B - Docetaxel Then Liposomal Doxorubicin
Started | 32 | 24
Completed | 32 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A -Liposomal Doxorubicin Then Docetaxel: Liposomal doxorubicin (Arm A)
  Liposomal doxorubicin 40 mg/m2 IV day 1 over one hour, repeated q 28 days thru peripheral vein or central venous access. This will define one cycle.
  Patients demonstrating progression on Liposomal Doxorubicin were eligible for cross over to treatment on Docetaxel, provided the patient still met the eligibility laboratory and performance status criteria.
- Arm B - Docetaxel Then Liposomal Doxorubicin: Weekly docetaxel 36 mg/m2 IV over 30 minutes on days 1, 8 and 15 followed by one week rest, administered on a q 28 day cycle. This dosing schedule will define one cycle.
  Patients demonstrating progression on Docetaxel were eligible for cross over to treatment on Liposomal Doxorubicin, provided the patient still met the eligibility laboratory and performance status criteria.
- Total: Total of all reporting groups
Arm/Group | Arm A -Liposomal Doxorubicin Then Docetaxel | Arm B - Docetaxel Then Liposomal Doxorubicin | Total
Number analyzed (Participants) | 50 | 52 | 102
Age Continuous [Median (Full Range); unit: years] | 62 [31 to 87] | 62 [31 to 87] | 62 [31 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 52 | 102
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: ORR is defined as the percentage of patients who exhibit a Complete Response (CR) or Partial Response (PR). Complete Response is the total disappearance of clinically and radiologically detectable disease for at least 4 weeks. Partial Response is at least a 50% reduction of all measurable lesions as measured by the product of the perpendicular diameters of the greatest dimensions of tumor size, with no new lesions appearing for at least four weeks.
Time Frame: 18 Months
Population: Patients who were removed from treatment before evaluation were not included in analysis
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A -Liposomal Doxorubicin Then Docetaxel | Arm B - Docetaxel Then Liposomal Doxorubicin
Number analyzed (Participants) | 42 | 44
percentage of patients | 28 [16 to 42] | 31 [18 to 45]

2. Secondary Outcome: Progression Free Survival (PFS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease.
Description: PFS was defined as the interval from first study treatment until the date that the first progression of breast cancer was documented, or death occurred.
Time Frame: 18 Months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A -Liposomal Doxorubicin Then Docetaxel | Arm B - Docetaxel Then Liposomal Doxorubicin
Number analyzed (Participants) | 48 | 44
months | 6.5 [3.6 to 9.5] | 5.5 [4.9 to 9.6]

ADVERSE EVENTS:
Groups:
- Arm A - Liposomal Doxorubicin Then Docetaxel: Liposomal doxorubicin 40 mg/m2 IV day 1 over one hour, repeated q28 days thru peripheral vein or central venous access. This will define one cycle. Patients demonstrating progression on Liposomal Doxorubicin were eligible for crossover to treatment on Docetaxel, provided patient still met the eligibility lab and performance status criteria.
- Arm B - Docetaxel Then Liposomal Doxorubicin: Weekly docetaxel 36 mg/m2 IV over 30 minutes on days 1, 8, and 15 followed by one week rest, administered on an every 28 day cycle. This dosing schedule will define one cycle. Patients demonstrating progression on Docetaxel were eligible for cross over to treatment on Liposomal Doxorubicin, provided patient still met the eligibility laboratory and performance status criteria.
Arm/Group | Arm A - Liposomal Doxorubicin Then Docetaxel | Arm B - Docetaxel Then Liposomal Doxorubicin
Serious Adverse Events (participants affected / at risk) | 18/50 | 22/52
Other Adverse Events (participants affected / at risk) | 21/50 | 35/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Liposomal Doxorubicin Then Docetaxel (N=50) | Arm B - Docetaxel Then Liposomal Doxorubicin (N=52)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Failure to Thrive (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subtrochanteric Fracture
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Liver Dysfunction (Hepatobiliary disorders) | 1 (1) | 1 (1) — Jaundice
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain - Abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage - GI (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Superior Vena Cava Syndome (Vascular disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain - Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Diverticular Abscess (Gastrointestinal disorders) | 1 (1) | 0 (0)
CNS Ischemia (Nervous system disorders) | 1 (1) | 0 (0) — Cerebrovascular Accident (CVA)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Liposomal Doxorubicin Then Docetaxel (N=50) | Arm B - Docetaxel Then Liposomal Doxorubicin (N=52)
Neutrophils (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Fatigue (General disorders) | 3 (3) | 13 (13)
Mucositis/Stomatitis (Gastrointestinal disorders) | 4 (4) | 3 (3)
Hand-Foot (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2) | 6 (6)
Arthralgia/Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Edema (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Hypotension (Cardiac disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.